CLINICAL TRIAL: NCT06745596
Title: Anterior Segment Changes After Phacoemulsification in Cataractous Eyes with Shallow Anterior Chamber with and Without Limited Anterior Pars Plana Vitrectomy
Brief Title: Anterior Segment Changes After Phacoemulsification in Cataractous Eyes with Shallow Anterior Chamber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #467/24-June-2024.; Zagazig university (Other: Zagazig university)
Record Dates: First submitted 2024-12-06; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Cataract
Keywords: Limited anterior pars plana vitrectomy
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: 24 eyes were operated on and divided into two groups. Twelve eyes underwent combined approach and the other 12 eyes have undergone phacoemulsification only
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cataract with limited anterior pars plana vitrectomy (Active Comparator): group I included twelve patients who underwent phacoemulsification combined with limited anterior pars plana vitrectomy
  Interventions: Procedure: cataract surgery 1
- Cataract without limited anterior pars plana vitrectomy (Active Comparator): group II included twelve patients that underwent phacoemulsification only
  Interventions: Procedure: cataract surgery 2

INTERVENTIONS:
Procedure: cataract surgery 1 — Cataract with limited anterior pars plana vitrectomy
  Arms: Cataract with limited anterior pars plana vitrectomy
Procedure: cataract surgery 2 — cataract without limited anterior pars plana vitrectomy
  Arms: Cataract without limited anterior pars plana vitrectomy

SUMMARY:
Phacoemulsification in shallow anterior chamber is considered to be more hazardous regarding risk of intraoperative and postoperative complications. Limited anterior pars plana vitrectomy can be combined with phacoemulsification to deepen the anterior chamber and facilitate surgical steps

DETAILED DESCRIPTION:
Phacoemulsification in shallow anterior chamber is considered to be more hazardous regarding risk of intraoperative and postoperative complications. Limited anterior pars plana vitrectomy can be combined with phacoemulsification to deepen the anterior chamber and facilitate surgical steps. This study aimed to compare the efficacy of combined phacoemulsification with limited pars plana vitrectomy versus phacoemulsification alone in cases with shallow anterior chamber.

Methods: 24 eyes were operated on and divided into two groups. Twelve eyes underwent combined approach and the other 12 eyes have undergone phacoemulsification only.

ELIGIBILITY:
Inclusion criteria:

* Anterior chamber depth of less than 2.8 mm associated with cataract

Exclusion Criteria:

* Mature cataract
* History of previous ocular surgery
* Posterior segment pathology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Central corneal thickness in micrometers. | 6 months
  Central corneal thickness in both groups measured by anterior segment OCT

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Mohammad Gamal Mohammad Gamal, MBBCh, Study Director — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No